CLINICAL TRIAL: NCT01903356
Title: A Regulatory Requirement Non Interventional Study to Monitor the Safety and Effectiveness of Trajenta Duo® (Linagliptin/Metformin HCl, 2.5 mg/500 mg, 2.5 mg/850 mg and 2.5 mg/1000 mg, b.i.d) in Korean Patients With Type 2 Diabetes Mellitus
Brief Title: A Regulatory Requirement Non Interventional Study to Monitor Safety and Effectiveness of Trajenta Duo in Type 2 Diabetes Patients in Korea
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1288.22
Record Dates: First submitted 2013-07-16; First posted 2013-07-19 (Estimated); Results first posted 2018-12-21 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with T2DM
  Interventions: Drug: Trajenta duo

INTERVENTIONS:
Drug: Trajenta duo — Linagliptin and Metformin

SUMMARY:
The primary objective of this study is to monitor the safety profile of Trajenta Duo in Korean patients with type 2 diabetes mellitus (T2DM) in a routine clinical setting.

DETAILED DESCRIPTION:
Study Design:

Post Marketed Study- Observational study

ELIGIBILITY:
Inclusion criteria:

Potential subjets must meet all of the following inclusion criteria to enter this trial:

1. No previous exposure to Trajenta, Trajenta Duo
2. Should have been started on Trajenta Duo in accordance with the approved label in Korea
3. No current participation in clinical trials
4. No metformin is inappropriate due to contraindications
5. Must sign on the data release consent form

Exclusion criteria:

Individuals with any of the following characteristics will not be able to enter this study:

1. Previous exposure to Trajenta, Trajenta Duo
2. Current participation in clinical trials
3. Patients for whom metformin is inappropriate due to contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean patients with T2DM
Sampling Method: Probability Sample
Enrollment: 724 (Actual)
Dates: Start 2013-07-11 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Multiple Locations, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an observational study in patients with type 2 diabetes mellitus who had been administered with TrajentaDuo® Tablets. The Case Report Forms of 724 subjects investigated by 15 investigators at 14 hospitals were retrieved from November 15, 2012 up to September 13, 2017.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that all subjects met all inclusion/exclusion criteria. Subjects were not to be enrolled in the study if any one of the specific entry criteria were violated.
Groups:
- TrajentaDuo® Tablet: Patients with type 2 diabetes mellitus (T2DM) were administered with oral dose of TrajentaDuo® (Linagliptin/Metformin hydrochloride (HCl) fixed dose combination, 2.5 mg/500 mg, 2.5 mg/850 mg or 2.5 mg/1000 mg, twice daily) Tablet
Period: Overall Study
Arm/Group | TrajentaDuo® Tablet
Started | 724
Completed | 709
Not Completed | 15
Not completed — Lost to Follow-up | 7
Not completed — Violated inclusion/exclusion criteria | 5
Not completed — Violated the dosage and administration | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: This analysis set included all subjects except subjects violating inclusion/exclusion criteria, dosage adminstration or were lost to follow up.
Arm/Group | TrajentaDuo® Tablet
Number analyzed (Participants) | 709
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age of all patients enrolled in the study Population: Safety Analysis Set: This analysis set included all subjects except subjects violating inclusion/exclusion criteria, dosage adminstration or were lost to follow up.
  Years | 62.04 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender distribution of all patients enrolled in the study Population: Safety Analysis Set: This analysis set included all subjects except subjects violating inclusion/exclusion criteria, dosage adminstration or were lost to follow up.
  Participants
    Female | 358
    Male | 351
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hemoglobin A1c (HbA1c) at baseline [Mean (Standard Deviation); unit: Percentage of HbA1c (%)] — HbA1c values measured at baseline in percent. HbA1c is a form of hemoglobin, a blood pigment that carries oxygen, which is bound to glucose. The term HbA1c also refers to glycated hemoglobin. High levels of HbA1c (Normal range is less than 6%) indicate poorer control of diabetes than level in normal range. Population: Effectiveness Analysis Set: This analysis set included all subjects from safety analysis set for whom HbA1c was recorded before administration of treatment and at least once after treatment for at least 10 weeks.
  Percentage of HbA1c (%)
    number analyzed (Participants) | 481
    (all) | 7.78 (1.35)

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) After 24 Weeks of Treatment.
Description: This outcome has measured difference between HbA1c values from baseline to 24 weeks post treatment. The term 'baseline' refers to the last observation prior to the administration of any study medication. HbA1c is a form of hemoglobin, a blood pigment that carries oxygen, which is bound to glucose. The term HbA1c also refers to glycated hemoglobin. High levels of HbA1c (Normal range is less than 6%) indicate poorer control of diabetes than level in normal range.
Time Frame: Baseline and Week 24
Population: Effectiveness Analysis Set: This analysis set included all subjects from safety analysis set for whom HbA1c was recorded before administration of treatment and at least once after treatment for at least 10 weeks.
Measure: Mean (Standard Deviation); unit: Percentage (%) of HbA1c
Arm/Group | TrajentaDuo® Tablet
Number analyzed (Participants) | 481
Percentage (%) of HbA1c | -0.75 (1.48)
Statistical Analysis 1: Comparison: TrajentaDuo® Tablet; Comparison of % of HbA1c before and 24 weeks after administration of TrajentaDuo® Tablet treatment; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test has been used for this analysis; The difference considered in the analysis is HbA1c values after drug administration minus HbA1c values before drug administration

2. Secondary Outcome: Target Effectiveness Response Rate
Description: Occurrence of treatment to target effectiveness response is an HbA1c under treatment of < 6.5% after 24 weeks of treatment. This outcome measures percentage of patients achieving HbA1c < 6.5% after 24 weeks.
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients (%)
Arm/Group | TrajentaDuo® Tablet
Number analyzed (Participants) | 481
Percentage of Patients (%) | 33.06

3. Secondary Outcome: Relative Effectiveness Response Rate
Description: Occurrence of relative effectiveness response. This outcome measures percentage of patients for which HbA1c has reduced by at least 0.5% after 24 weeks.
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of patients (%)
Arm/Group | TrajentaDuo® Tablet
Number analyzed (Participants) | 481
Percentage of patients (%) | 46.78

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) After 24 Weeks of Treatment.
Description: This outcome has measured difference between Fasting Plasma Glucose (FPG) values from baseline to 24 weeks post treatment. The term 'baseline' refers to the last observation prior to the administration of any study medication.
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milligram/deciLitre (mg/dL)
Arm/Group | TrajentaDuo® Tablet
Number analyzed (Participants) | 481
Milligram/deciLitre (mg/dL) | -17.12 (52.60)
Statistical Analysis 1: Comparison: TrajentaDuo® Tablet; Comparison of FPG before and 24 weeks after administration of TrajentaDuo® Tablet treatment; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test has been used for this analysis; The difference considered in the analysis is FPG values after drug administration minus FPG values before drug administration

5. Primary Outcome: Incidence Rate of Adverse Events (AE)
Description: The incidence rate is the number of new cases per population at risk in a given time period. The incidence rate was calculated in patients who take at least one Trajenta Duo
Time Frame: Up to 26 weeks
Population: as for baseline characteristics
Measure: Number; unit: Percentage of patients (%)
Arm/Group | TrajentaDuo® Tablet
Number analyzed (Participants) | 709
Percentage of patients (%) | 11.99

ADVERSE EVENTS:
Time Frame: From first drug administration until 24 weeks of treatment administration, up to approximately 252 weeks after last visit.
Description: An adverse event (AE) is defined as any untoward medical occurrence, including an exacerbation of a pre-existing condition, in a patient in a clinical investigation who received a pharmaceutical product. The event does not necessarily have to have a causal relationship with this treatment. All reported adverse events including hypoglycemic events in patients who take at least one dose of Trajenta Duo® were noted.
Arm/Group | TrajentaDuo® Tablet
All-Cause Mortality (participants affected / at risk) | 0/709
Serious Adverse Events (participants affected / at risk) | 15/709
Other Adverse Events (participants affected / at risk) | 0/709
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TrajentaDuo® Tablet (N=709)
Angina pectoris (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Mediastinitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Vitreous haemorrhage (Eye disorders) | 1
Pyrexia (General disorders) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT01903356/Prot_SAP_000.pdf